CLINICAL TRIAL: NCT06205238
Title: The Impact of Domiciliary Versus 'Hub' Based Comprehensive Geriatric Assessment on Clinical and Process Outcomes Among Older Adults Attending Community Specialist Teams: a Randomised Controlled Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRB RL2020-010
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Frailty; Comprehensive Geriatric Assessment; Older Adults; Domiciliary Care
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to group allocation to reduce detection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Domiciliary CGA (Experimental): The intervention will consist of domiciliary CGA including nursing, medical and allied health assessment and intervention for frail older adults over age 75 who are discharged the ED or referred urgently from their GP and referred to the CST in Limerick. The bulk of this intervention will be delivered in the patient's own home. Each participant will be required to attend the hub for their medical review where they will access specialist geriatric medical expertise. A domiciliary visit to the older person within 24-48 hours of referral from the ED or within 24-48 hours of triage of GP referral by a member of the multidisciplinary team. This person will act as the case coordinator. During this visit, there will be a detailed assessment of the older adult. Referrals will be made for domiciliary care to the appropriate healthcare professionals based on patient. The template proposed by Ellis et al. (2017) will be used to characterise the components of the CGA intervention.
  Interventions: Other: CGA
- Hub-based CGA (Active Comparator): The intervention will consist of CGA as defined above, including nursing, medical and allied health assessment and intervention for frail older adults over age 75 who are discharged the ED or referred urgently from their General Practitioner and referred to the CST in Limerick and will be seen in the Out-patient CST setting.
  Interventions: Other: CGA

INTERVENTIONS:
Other: CGA — CGA is defined as a "multidimensional interdisciplinary diagnostic process focused on determining a frail elderly person's medical, psychological and functional capability in order to develop a coordinated and integrated plan for treatment and long term follow up".

SUMMARY:
The investigators plan to implement a randomised controlled trial to examine the impact of domiciliary (home based) versus 'hub-based' Comprehensive Geriatric Assessment (CGA) on clinical and process outcomes among older adults referred to a community specialist team for older persons in the Mid-West region of Ireland. The population of interest is older adults who are discharged directly from the Emergency Department or referred urgently from their General Practitioner. The outcomes of interest focus on those that matter most to older adults as well as clinical and process measures of care.

DETAILED DESCRIPTION:
CGA is defined as a "multidimensional interdisciplinary diagnostic process focused on determining a frail elderly person's medical, psychological and functional capability in order to develop a coordinated and integrated plan for treatment and long term follow up" (1). The CST hub in Limerick provides a rapid, single point of access to an outpatient specialist geriatrician and allied health professional assessment. The bulk of this therapy is delivered in each of the hubs. This is considered 'usual' or routine care for the purposes of this trial.

The intervention will consist of domiciliary multidisciplinary CGA and intervention including nursing, medical and allied health assessment and intervention for frail older adults over age 75 who are discharged from the ED, or referred urgently from their General Practitioner and referred to the CST in Limerick. The bulk of this intervention will be delivered in the patient's own home. Each participant will be required to attend the hub for their medical review where they will access specialist geriatric medical expertise. A domiciliary visit to the older person within 24-48 hours of referral from the ED or within 24-48 hours of triage of GP referral by a member of the multidisciplinary team will be carried out. This person will act as the case coordinator for the duration of the intervention. During this visit, there will be a detailed assessment of the older adult. The assessment will include but not be limited to a falls assessment, assessment of mobility and stairs, transfer, personal care, activities of daily living (ADLs), social supports, cognition, lying & standing blood pressures and nutritional assessment. Referrals will be made for domiciliary care to the appropriate healthcare professionals (nursing, OT, physiotherapy, dietetics etc) based on the findings of this holistic assessment. Interventions prescribed will be individualised based on patient needs. The investigators will use the template proposed by Ellis et al. (2017) to characterise the components of the CGA intervention.

The trial will assess the benefits of this domiciliary model of care on outcomes including the following: function, quality of life, patient satisfaction, primary and secondary healthcare use, nursing home admission, mortality and cost-effectiveness. Baseline measurement will be taken at their index visit with follow-up at six weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the CST hub from a General Practitioner (urgent referral) or from the ED at University Hospital Limerick.

All of criteria 1-5 must be met

1. 75 years and over
2. Evidence of frailty, scoring between 4 and 6 on the Rockwood Clinical Frailty Scale (pre-frail, mildly frail or moderately frail)
3. Resides within CHO 3 and the catchment area of the relevant ICPOP hub
4. Patient has been assessed in-person by the referrer
5. Patient has not had MDT input within the last three months (excluding OPTIMEND team)

   And any one of criteria 6-10 must be met:
6. Fall within the last month unrelated to acute cardiac or neurological cause & no previous falls assessment
7. Increased dependency or increased carer burden in the last month
8. A deterioration in swallow in the last month including symptoms of recurrent chest infections, weight loss, coughing when eating/drinking, self-modifying diet secondary to difficulties
9. Adverse drug reaction within the last month excluding allergic reaction Referred from ED/AMU following review by consultant in Emergency Medicine, Acute Medicine, Geriatric Medicine, General Medicine or Frailty at the Front Door team

Exclusion Criteria:

* Present with an acute neurological or cardiovascular event
* Are more appropriate to an alternative care pathway or service e.g. primary care or geriatric medicine clinic
* Present with injuries, unless the injury has already been appropriately managed,
* Are experiencing an acute medical illness requiring treatment in an acute hospital setting
* If care is being provided by other health care professionals at the time of referral and it is apparent that they are working to meet goals aligned with the current service
* They require investigation or treatment not available in the relevant ICPOP hub (unless these investigations are already being arranged elsewhere)
* They have had MDT input in the last three months
* Have confirmed or suspected Covid-19 infection
* Or other exclusions at the discretion of the integrated care team based on clinical expertise and available resource.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional status | Baseline
  Barthel Index
Functional status | 6-weeks
  Barthel Index
Functional status | 6-months
  Barthel Index
Functional status | 12-months
  Barthel Index

SECONDARY OUTCOMES:
Unplanned ED revisit | Baseline
  Process measure for hospital data base
Unplanned ED revisit | 6-weeks
  Process measure for hospital data base
Unplanned ED revisit | 6-months
  Process measure for hospital data base
Unplanned hospitalisation | Baseline
  Process measure for hospital data base
Unplanned hospitalisation | 6-weeks
  Process measure for hospital data base
Unplanned hospitalisation | 6-months
  Process measure for hospital data base
Nursing Home admission | 6-weeks
  Process measure
Nursing Home admission | 6-months
  Process measure
Mortality | 6-weeks
  The number of participants who died following their index visit
Mortality | 6-months
  The number of participants who died following their index visit
Health related quality of life (HRQOL) | Baseline
  EuroQoL-5D-5L
Health related quality of life (HRQOL) | 6-weeks
  EuroQoL-5D-5L
Health related quality of life (HRQOL) | 6-months
  EuroQoL-5D-5L
Patient satisfaction with care | 6-weeks
  Patient Assessment of Integrated Elderly Care Questionnaire
Patient satisfaction with care | 6-months
  Patient Assessment of Integrated Elderly Care Questionnaire
Primary healthcare use (outside of community specialist team for older persons) | 6-weeks
  Process measure
Primary healthcare use (outside of community specialist team for older persons) | 6-months
  Process measure
Number of healthcare professional encounters by the community specialist team for older persons | 6-weeks
  Process measure
Number of healthcare professional encounters by the community specialist team for older persons | 6-months
  Process measure
Unplanned ED revisit | 12-months
  Process measure for hospital data base
Unplanned hospitalisation | 12-months
  Process measure for hospital data base
Nursing Home admission | 12-months
  Process measure
Mortality | 12-months
  The number of participants who died following their index visit
Health related quality of life (HRQOL) | 12-months
  EuroQoL-5D-5L
Primary healthcare use (outside of community specialist team for older persons) | 12-months
  Process measure

CONTACTS AND LOCATIONS:
Locations (1):
- Community Specialist Team Hub, Limerick, Munster, Ireland